CLINICAL TRIAL: NCT03859388
Title: Use of Donor-Derived Cell-Free DNA to Characterize Response to Therapy With Tocilizumab for Chronic Antibody-Mediated Rejection in Kidney Transplantation
Brief Title: Longitudinal Changes in Donor-Derived Cell-Free DNA With Tocilizumab Treatment for Chronic Antibody-Mediated Rejection
Status: Active, not recruiting | Type: Observational
Sponsor: Cedars-Sinai Medical Center (Other)
Responsible Party: Principal Investigator, Edmund Huang, Health Sciences Associate Professor of Medicine, Cedars-Sinai Medical Center
Other Study IDs: Pro00053105
Record Dates: First submitted 2019-02-25; First posted 2019-03-01 (Actual); Last update posted 2025-04-24 (Actual); Status verified 2025-04

CONDITIONS: Rejection Chronic Renal; Kidney Transplant Rejection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Chronic ABMR: Single arm; patients with chronic ABMR diagnosed by Banff 2017 criteria and recommended for monthly treatment with tocilizumab will undergo monthly testing for donor-derived cell-free DNA (Allosure) and then have a follow-up biopsy after six monthly infusions of tocilizumab

SUMMARY:
Our group recently reported that tocilizumab, a humanized monoclonal antibody against the IL-6 receptor, may be effective when administered monthly to patients with chronic antibody-mediated rejection (ABMR). The current paradigm to assess response to therapy involves serial monitoring for donor-specific antibodies, measurement of kidney function with creatinine, and periodic kidney transplant biopsies to survey for histologic findings indicative of ongoing ABMR.

A new non-invasive blood test, donor-derived cell-free DNA (Allosure) has recently reported to have a high degree of discrimination for rejection and may be used to assess the likelihood of rejection. It has not been tested to see if it can be used to assess treatment response for rejection.

This study will assess longitudinal changes in donor-derived cell-free DNA measurements in response to monthly therapy with tocilizumab for chronic ABMR and correlate these measurements to histologic changes on a follow-up kidney transplant biopsy.

DETAILED DESCRIPTION:
Chronic antibody-mediated rejection (ABMR) is now recognized as the leading cause of late kidney transplant failure (1). A number of new immunosuppressive medications have been introduced to the field of kidney transplantation over the last twenty years, leading to a reduction in early acute rejection rates (2). However, long-term graft survival has not improved, primarily because of failure to make a timely diagnosis of chronic ABMR and a lack of effective therapeutic options. To date, treatment options for chronic ABMR are limited and include intravenous immunoglobulin (IVIg), rituximab, and plasmapheresis. These agents are effective for treatment of acute ABMR; however, they are generally ineffective in sustaining kidney function and prolonging graft survival in chronic ABMR.

Interleukin-6 (IL-6) blockade has emerged as a promising therapy for chronic ABMR. Our group recently reported that tocilizumab, a humanized monoclonal antibody against the IL-6 receptor, administered monthly to patients with chronic ABMR is associated with a reduction in donor specific antibodies (DSA), stabilization of renal function, improvement in histologic features of chronic ABMR, and excellent patient and graft survival up to six years (3).

The diagnostic criteria for antibody-mediated rejection in kidney transplantation requires serologic evidence of donor-specific antibodies to human leukocyte antigen (HLA) or other antigens in conjunction with histologic findings of ABMR on biopsy for a definitive diagnosis of ABMR (4). The criteria recognize that the mere presence of DSA alone is not sufficient to classify a patient as having ABMR, as has been described previously (5). Among patients treated for ABMR, a reduction in DSA is associated with a favorable response but is only observed in a small percentage of treated patients (6). Among patients with chronic ABMR who are treated, there is a subset with persistence of high titer DSA, yet stable renal function and resolution of active lesions of ABMR on follow-up kidney biopsy. Although these patients may not warrant continuing therapy with tocilizumab, they cannot be distinguished from patients with persistently active ABMR without undergoing an additional allograft biopsy. A non-invasive test for ABMR is preferred, as allograft biopsies are invasive, resource-intensive, carry a risk of bleeding, and are time-consuming for the patient. If validated, non-invasive testing for ABMR can be useful for monitoring for a treatment response and may help guide therapy for ABMR.

Because donor-derived cell-free DNA (Allosure) is predictive of rejection n kidney transplantation, longitudinal changes in the percentage of donor-derived cell free DNA detected in plasma of kidney transplant recipients with chronic ABMR may correlate with a histologic and clinical response to treatment. The primary objective is to assess whether longitudinal changes in donor-derived cell-free DNA correlate with histologic and clinical response to treatment with tocilizumab for chronic ABMR. The secondary objectives are to assess the test performance of donor-derived cell-free DNA measured against histologic findings on biopsy, provide molecular evidence for response to tocilizumab therapy, and to describe the time course of treatment effect of tocilizumab in chronic ABMR.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* Enrolled within six months of biopsy-proven evidence of chronic active ABMR defined by Banff 2017 diagnostic criteria
* Evidence of DSA detected in the blood within 6 months prior to consent.
* Able to understand and provide informed consent.

Exclusion Criteria:

* Known contraindications for therapy with tocilizumab:
* Hypersensitivity
* Elevated liver enzymes
* Patients at risk for GI perforation
* Absolute neutrophil count <500/mm3
* Platelet count <50,000/mm3
* Active infection
* Contraindications for kidney transplant biopsy, including bleeding diathesis or technical/anatomical infeasibility for biopsy.
* Contraindications to donor-derived cell-free DNA (AlloSure) testing:
* Recipient of multiple transplanted organs.
* Recipient of a transplant from an identical twin.
* Pregnant
* Under the age of 18.
* Less than two weeks post-transplant.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult recipients of a kidney transplant alone who have chronic active ABMR on kidney transplant biopsy and are recommended for treatment with tocilizumab
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2019-03-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in the percentage of donor-derived cell-free DNA | 12 months
  Change in % donor-derived cell-free DNA/month

SECONDARY OUTCOMES:
Difference in Change in Donor-Derived Cell-Free DNA Between Responders and Non-Responders | 6 months
  Difference in the mean delta of donor-derived cell-free DNA from baseline to six months among histologic responders and non-responders (paired t-test)
Change in estimated glomerular filtration rate (GFR) | 12 months
  Change in estimated glomerular filtration rate (GFR) measured by the Chronic Kidney Disease Epidemiology Collaboration (CKD-EPI) equation over 12 months from initiation of tocilizumab treatment (linear mixed effects model)
Change in glomerulitis histology score with treatment | 6 months
  Change in histologic features of ABMR before and after 6 months of treatment with tocilizumab (paired t-test; g-score)
Change in peritubular capillaritis histology score with treatment | 6 months
  Change in histologic features of ABMR before and after 6 months of treatment with tocilizumab (paired t-test; ptc-score)
Change in C4d score with treatment | 6 months
  Change in histologic features of ABMR before and after 6 months of treatment with tocilizumab (paired t-test; C4d-score)
Change in glomerular double contours score with treatment | 6 months
  Change in histologic features of ABMR before and after 6 months of treatment with tocilizumab (paired t-test; cg-score)
Change in interstitial fibrosis score with treatment | 6 months
  Change in histologic features of ABMR before and after 6 months of treatment with tocilizumab (paired t-test; ci-score)
Change in tubular atrophy score with treatment | 6 months
  Change in histologic features of ABMR before and after 6 months of treatment with tocilizumab (paired t-test; ct-score)

CONTACTS AND LOCATIONS:
Overall Officials: Edmund Huang, M.D., Principal Investigator — Cedars-Sinai Medical Center
Locations (1):
- Cedars-Sinai Medical Center, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sellares J, de Freitas DG, Mengel M, Reeve J, Einecke G, Sis B, Hidalgo LG, Famulski K, Matas A, Halloran PF. Understanding the causes of kidney transplant failure: the dominant role of antibody-mediated rejection and nonadherence. Am J Transplant. 2012 Feb;12(2):388-99. doi: 10.1111/j.1600-6143.2011.03840.x. Epub 2011 Nov 14. PMID 22081892
- [Background] Meier-Kriesche HU, Schold JD, Srinivas TR, Kaplan B. Lack of improvement in renal allograft survival despite a marked decrease in acute rejection rates over the most recent era. Am J Transplant. 2004 Mar;4(3):378-83. doi: 10.1111/j.1600-6143.2004.00332.x. PMID 14961990
- [Background] Choi J, Aubert O, Vo A, Loupy A, Haas M, Puliyanda D, Kim I, Louie S, Kang A, Peng A, Kahwaji J, Reinsmoen N, Toyoda M, Jordan SC. Assessment of Tocilizumab (Anti-Interleukin-6 Receptor Monoclonal) as a Potential Treatment for Chronic Antibody-Mediated Rejection and Transplant Glomerulopathy in HLA-Sensitized Renal Allograft Recipients. Am J Transplant. 2017 Sep;17(9):2381-2389. doi: 10.1111/ajt.14228. Epub 2017 Mar 10. PMID 28199785
- [Background] Haas M. The Revised (2013) Banff Classification for Antibody-Mediated Rejection of Renal Allografts: Update, Difficulties, and Future Considerations. Am J Transplant. 2016 May;16(5):1352-7. doi: 10.1111/ajt.13661. Epub 2016 Feb 4. PMID 26696524
- [Background] Eskandary F, Regele H, Baumann L, Bond G, Kozakowski N, Wahrmann M, Hidalgo LG, Haslacher H, Kaltenecker CC, Aretin MB, Oberbauer R, Posch M, Staudenherz A, Handisurya A, Reeve J, Halloran PF, Bohmig GA. A Randomized Trial of Bortezomib in Late Antibody-Mediated Kidney Transplant Rejection. J Am Soc Nephrol. 2018 Feb;29(2):591-605. doi: 10.1681/ASN.2017070818. Epub 2017 Dec 14. PMID 29242250
- [Background] Haas M, Mirocha J, Reinsmoen NL, Vo AA, Choi J, Kahwaji JM, Peng A, Villicana R, Jordan SC. Differences in pathologic features and graft outcomes in antibody-mediated rejection of renal allografts due to persistent/recurrent versus de novo donor-specific antibodies. Kidney Int. 2017 Mar;91(3):729-737. doi: 10.1016/j.kint.2016.10.040. Epub 2017 Jan 16. PMID 28104301